CLINICAL TRIAL: NCT01655108
Title: BLIND RANDOMIZED COMPARATIVE STUDY TO EVALUATE THE EFFICACY AND SAFETY OF MESOTHERAPY MINOXIDIL HAIR WITH 0.5% / 2ML VERSUS PLACEBO IN THE TREATMENT OF FEMALE ANDROGENETIC ALOPECIA
Brief Title: Efficacy and Safety of Mesotherapy With Minoxidil 0.5%/2ml for Androgenetic Alopecia in Female Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Izelda Maria Carvalho Costa, Adjunct Professor, Brasilia University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUB-UnB TrichoGroup 1
Record Dates: First submitted 2012-07-24; First posted 2012-08-01 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Female Pattern Alopecia
Keywords: Androgenetic Alopecia; Mesotherapy; Minoxidil; Trichogram
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Placebo Comparator): After having been properly diagnostic as having androgenetic alopecia, through biopsy of the scalp, trichogram and trichoscopy and randomized in the placebo group, thirty women will be subjected to intradermal application (mesotherapy) of saline; ten sessions will be held at weekly intervals. Eight weeks after the last session will be repeated all the tests for comparison of results.
  Interventions: Drug: Saline
- Minoxidil 0.5% /2ml (Active Comparator): After having been properly diagnostic as having androgenetic alopecia, through biopsy of the scalp, trichogram and trichoscopy and randomized in the drug active group, thirty women will be subjected to intradermal application (mesotherapy) of minoxidil 0.5%/2ml; ten sessions will be held at weekly intervals. Eight weeks after the last session will be repeated all the tests for comparison of results.
  Interventions: Drug: Minoxidil

INTERVENTIONS:
Drug: Minoxidil — Minoxidil 0.5% /2ml intradermal injection in the scalp ( mesotherapy), weekly sessions, ten weeks
  Arms: Minoxidil 0.5% /2ml
Drug: Saline — Physiological saline solution 0.9% , intradermal injection in the scalp ( mesotherapy), weekly sessions, ten weeks
  Arms: Saline

SUMMARY:
This study aims to investigate the effectiveness and safety of mesotherapy for the treatment of female pattern alopecia.

* Sixty female subjects between 18 and 65 years diagnosed with female pattern hair loss will undergo mesotherapy sessions weekly for ten weeks.
* One group will receive 0.5%/2ml minoxidil application and a control group will receive application of placebo (saline 0.9%).
* Biopsy of the scalp, trichogram and trichoscopy (Fotofinder) will be performed before and 08 weeks after treatment as a method objective evaluation of the response

DETAILED DESCRIPTION:
This is a trial that aims to analyze the efficacy and safety of mesotherapy with minoxidil 0,5% versus placebo for androgenetic alopecia in female patients.

The patients and the investigators who analyzes complementary exams are blind.

* Clinical criteria, photo, 4mm biopsia, trichogram and trichoscopy are perfomed before patients are randomized into two arms :

  1. Group 1 (Placebo):

     30 patients who will have intradermal injections in the scalp of saline 0.9%
  2. Group 2 (Active Drug):

     30 patients who will receive intradermal injections in the scalp with minoxidil 0.5%/2ml

     Eight weeks after the last session patients will be recruited for repeat the exams and perform a self-assessment of both the effect on hair growth and the effect on hair loss.

ELIGIBILITY:
Inclusion Criteria:

* Women from 18 to 65 years old
* Androgenetic Alopecia (female pattern hair loss)

Exclusion Criteria:

* patients with alopecia areata or cicatricial alopecia
* pregnancy and breastfeeding
* have undergone any specific treatment in the last 06 months
* use of drugs with anti-androgenic properties
* patients with signs or symptoms of hyper-androgynism

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Increase in hair density | Sixteen weeks
  Six weeks after the last session of mesotherapy patients will be subjected to control examinations to evaluation of results. Scalp biopsy to determine the terminal-vellus ratio, trichogram to assess the percentage of anagen hair, telogen and dystrophic and Trichoscan will be performed to see if there was improvement in hair density

SECONDARY OUTCOMES:
Mesotherapy safety | six months
  In each session of mesotherapy, blood pressure and cardiac frequency at baseline and 10 min after application of the drug will be measured to assess the safety profile of the solution of minoxidil to 0.5% when injected intradermally.
  Any adverse effect reported will be recorded on specific clinical form

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Uzel, M.D, Principal Investigator — University of Brasilia; Izelda Costa, Ph.D, Study Director — University of Brasilia
Locations (1):
- University of Brasilia, Brasília, Federal District, Brazil